CLINICAL TRIAL: NCT03069729
Title: Thermal Screening for Early Diabetic Peripheral Neuropathy (DPN)
Status: Completed | Type: Observational
Sponsor: VisionQuest Biomedical LLC (Industry)
Collaborators: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: R43DK104578-01 (NIH)
Record Dates: First submitted 2017-02-16; First posted 2017-03-03 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Diabetic Neuropathies; Diabetic Foot; Diabetic Retinopathy
Keywords: screen
MeSH Terms: conditions — Diabetic Neuropathies; Diabetic Foot; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: non-diabetic; no intervention
  Interventions: Other: no intervention
- Diabetics without DPN: diabetics without DPN; no intervention
  Interventions: Other: no intervention
- Diabetics with DPN: diabetics with DPN; no intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This study evaluates s system intended to detect bio-markers of DPN. No interventions are involved in this non-invasive study.

SUMMARY:
The goal of this research is to develop better tools for diagnosing illness of the feet and legs of people who have diabetes. Investigators will use thermal videos of the foot to aid in the refinement of a system designed to detect signs of diabetic peripheral neuropathy (DPN). The team of investigators will also look at diabetic eye disease and how it might relate to diabetic foot disease.

DETAILED DESCRIPTION:
This study focuses on further development and testing of a microvascular functional imaging system, a computer-based system for screening thermal video images, designed to detect biomarkers of diabetic peripheral neuropathy (DPN). Additionally, severity levels of diabetic retinopathy (DR) will be compared with those of DPN.

All participants in this study will undergo foot exams, thermal imaging of the foot, and standard retinal imaging. These non-invasive assessments will be performed at an initial study visit. Some of the participants will be offered additional study visits. One of the additional visits involves a standard nerve conduction velocity assessment by a neurologist, the other involves a DPN exam by a podiatrist.

Portions of the study take place at University of New Mexico Health Sciences Center (UNM HSC). The research utilizes services of the Clinical Translational Science Center (CTSC).

The study is approved by University of New Mexico Health Sciences Center's Human Research Review Committee (HRRC), which coordinates and supports the activities of the three federally mandated Human Research Review Committees (HRRCs) responsible for reviewing and approving all human research.

ELIGIBILITY:
Inclusion Criteria:

• Must be non-diabetic or diagnosed as diabetic for at least 5 years

Exclusion Criteria:

history of chemotherapy

* surgery below the knee within the last 2 years
* fractures below the know within the last 2 years
* history of stroke
* body mass index (BMI) greater than 35
* history of heart failure
* peacemaker or implantable cardiovascular defibrillator
* high blood pressure (over 180/100)
* end-stage renal (kidney) disease or renal (kidney) transplant
* peripheral edema greater than 2+ (swelling of the feet or hands)
* diabetic foot ulcers
* foot sores
* Raynaud's phenomenon
* tobacco use within the last month.
* treatment with glucocorticoids, including:

  * beclomethasone
  * betamethasone
  * budesonide
  * cortisone
  * dexamethasone
  * hydrocortisone
  * methylprednisolone
  * prednisolone
  * prednisone
  * triamcinolone

Ages: 35 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of diabetic and non-diabetic individuals who are otherwise healthy.
Sampling Method: Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Pattern of thermal recovery | 24 months
  The thermal recovery pattern after cold provocation will be different for each group studied.

SECONDARY OUTCOMES:
Correlation of DPN severity levels and DR severity levels | 18 months
  Correlation between severity levels of DR and DPN will be determined.
  The severity level of DR will be assessed by qualified retinal image readers. Level of severity will be assigned, based on the International Clinical Diabetic Retinopathy Disease Severity Scale, into 5 levels:
  1. No apparent retinopathy
  2. Mild nonproliferative diabetic retinopathy
  3. Moderate nonproliferative diabetic retinopathy
  4. Severe nonproliferative diabetic retinopathy
  5. Proliferative diabetic retinopathy
  The severity of DPN will be graded by utilizing data from assessments from a DPN exam performed by an experienced podiatrist, Nerve Conduction Velocity (NCV) test performed by a neurologist, and assessments performed by technicians. Data utilized will include:
  * NVC results
  * Vibration threshold, reported in seconds
  * Monofilament test of protective sensation

CONTACTS AND LOCATIONS:
Overall Officials: Peter Soliz, PhD, Principal Investigator — VisionQuest Biomedical LLC
Locations (1):
- VisionQuest Biomedical LLC, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No